CLINICAL TRIAL: NCT04575636
Title: Magnetic Resonance Lymphography in Upper Extremity Lymphedema and Healthy Subjects
Brief Title: MRL in the Upper Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL72424.068.19
Record Dates: First submitted 2020-07-15; First posted 2020-10-05 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Lymphedema of Upper Limb

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymphedema patients (Other): MRL examination in lymphedema patients
  Interventions: Diagnostic Test: Magnetic Resonance Lymphography
- Healthy volunteers (Other): MRL examination in healthy volunteers
  Interventions: Diagnostic Test: Magnetic Resonance Lymphography

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Lymphography — Magnetic Resonance Lymphography using Siemens 3T MRI unit and Gadobutrol as a contrast agent to visualize the lymphatic system

SUMMARY:
Objective: The aim of this study is to examine the feasibility and applicability of the MRL protocol for the upper extremity in Maastricht University Medical Center, and to examine the differences of the lymphatic system between lymphedema patients and healthy volunteers.

Study design: An explorative study of an MRL protocol for the upper extremity in Maastricht University Medical Center+.

Study population: There are two study groups. The first group (n=10) consists of patients with secondary lymphedema in the upper extremity. The second group (n=10) consists of healthy volunteers.

Intervention (if applicable):

All participants will undergo an MRL examination with the same protocol, developed in a previous 'proof of principle' study, in the Maastricht University Medical Center+.

After localizer scans, a T2-weighted sequence is used. Then a T1-weighted sequence will be made before the injection of contrast. After the injection of the contrast agent a T1-weighted sequences of the upper and lower arm are performed alternately.

Main study parameters/endpoints:

The primary outcome is to determine the feasibility and applicability of the MRL protocol by evaluating the images of the upper extremity in patients with secondary lymphedema and healthy subjects.

The secondary outcome is to assess the value of MRL in staging lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* informed consent
* BMI < 30 kg/m2

Group A:

- Secondary lymphedema in the upper extremity

Group B:

- Healthy volunteers

Exclusion Criteria:

* Active skin infection/erysipelas in the arm.
* Known allergy for a contrast agent
* History of surgical intervention in the arm.
* Contraindications for MRI with contrast; pregnancy, metals, prostheses, renal insufficiency, claustrophobia
* Active cancer
* Distant metastases

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
feasiblity of Magentic Resonance Lymphography (MRL) of the arm by evaluating the MRL output images | 0.5 hours per participant
  Describing lymphatic vessel characteristics in terms of size, diameter and course, and lymphedema symptoms such as dermal backflow or obstruction

SECONDARY OUTCOMES:
lymphedema staging by evaluating the MRL output images | 0.5 hours per participant
  Describing lymphedema stage, based on lymphatic vessel charasteristics and lymphedema symptoms as found at primary outcome. This is compared with ISL (clinical) lymphedema stage and ICG lymphography stage.

CONTACTS AND LOCATIONS:
Locations (1):
- Scannexus, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No